CLINICAL TRIAL: NCT06936917
Title: Impact of Timing for Computed Tomography and Post-Resuscitation Care Sequence on Short-Term Outcomes in Out-of-Hospital Cardiac Arrest
Brief Title: Timing for Computed Tomography and Post-Resuscitation Care on Short-Term Outcomes in Out-of-Hospital Cardiac Arrest
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202409129RINC
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-12

CONDITIONS: Out of Hospital Cardiac Arrest; Computed Tomography
Keywords: Out-of-hospital cardiac arrest; Computed tomography; short-term outcome; resuscitation management; cardiopulmonary resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA with ROSC and receive CT: Patients who experienced out-of-hospital cardiac arrest, received resuscitative efforts in the emergency department, achieved return of spontaneous circulation (ROSC), and subsequently underwent computed tomography (CT) imaging, regardless of the anatomical region scanned.

SUMMARY:
This retrospective multicenter study investigates the association between the timing of computed tomography (CT) scans and short-term outcomes in adult non-traumatic out-of-hospital cardiac arrest (OHCA) patients who achieved return of spontaneous circulation (ROSC). The study includes cases from January 1, 2016, to August 31, 2024, across six branches of National Taiwan University Hospital. Data collected include demographics, Utstein variables, emergency department (ED) interventions and their timing. Primary outcomes are survival to admission, and 1-day, 3-day, and 7-day survival. Secondary outcomes focus on the timing and sequence of CT imaging and other interventions in relation to short-term prognosis and ED length of stay. The study aims to explore whether earlier CT utilization can improve outcomes in the post-resuscitation phase of care.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) patients with return of spontaneous circulation (ROSC) would suffer from an inflammatory response in the body due to hypoxia and subsequent reperfusion injury, known as post-cardiac arrest syndrome (PCAS). Prompt interventions were crucial during this phase at the emergency department. Typically , these patients require rapid computed tomography (CT) scans. CT scans of different body parts aid in diagnosing serious infections (e.g., pneumonia, perforated peptic ulcer) and vascular emergencies (e.g., stroke, intracranial hemorrhage, aortic dissection, aneurysm, pulmonary embolism), enabling timely specialist intervention, catheterization, or surgery. Patients with traumatic cardiac arrest also require CT scans to identify the mechanism of fatal injuries and assess the current injury status.

Theoretically, the ED team would prefer to perform CT scans as quickly as possible after resuscitation. However, PCAS can result in unstable vital signs, and transporting unstable patients to the CT room, with limited resuscitation equipment, carries the risk of recurrent cardiac arrest. As a result, the patient's vitals are stabilized at ED before receiving the CT scan. However, delaying the scan also impedes diagnosis and treatment, prolonging the patient's unstable condition and creating a vicious cycle. Currently, there is no consensus or standard regarding the optimal timing for CT scans after resuscitation, with most literature focusing on brain CT scans. Thus, whether the timing and prioritization of CT scans can break this vicious cycle remains an area requiring further research.

This retrospective study is part of a sequential research effort by our team. We plan to include non-traumatic adult OHCA patients from January 2016 to August 2024 (2016/01/01 to 2024/08/31). The patient population will be drawn from NTU Hospital and its affiliated branches (Hsinchu, Biomedical, and Zhudong) and NTU Yunlin Branch (Huwei and Douliu), covering six hospital areas across three hospitals. Study variables include basic demographics, Utstein Style OHCA registry variables, ED interventions and their timing. Primary outcomes include survival to hospital admission, 1-day, 3-day, and 7-day survival rates. Secondary outcomes will examine the timing of CT scans, the sequence of other interventions, and their relationship to short-term survival and ED length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 years or older.
2. Patients who experienced out-of-hospital cardiac arrest (OHCA), received resuscitative efforts in the emergency department, achieved return of spontaneous circulation (ROSC), and subsequently underwent computed tomography (CT) imaging (regardless of the anatomical region scanned).

Exclusion Criteria:

1. Patients with cardiac arrest due to traumatic causes (traumatic OHCA).
2. Patients who were transferred to non-NTUH-affiliated hospitals for post-resuscitation care.
3. Patients whose prognosis could not be determined from medical records.
4. Patients with incomplete, missing, or otherwise restricted medical records that limited data accessibility or review.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OHCA and ROSC
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2027-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Short-term outcomes (1-day, 3-day, and 7-day in-hospital survival) | 24, 72, and 168 hours following hospital admission from ED
  Defined as survival at 24, 72, and 168 hours, respectively, following hospital admission.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branch KRH, Gatewood MO, Kudenchuk PJ, Maynard C, Sayre MR, Carlbom DJ, Edwards RM, Counts CR, Probstfield JL, Brusen R, Johnson N, Gunn ML. Diagnostic yield, safety, and outcomes of Head-to-pelvis sudden death CT imaging in post arrest care: The CT FIRST cohort study. Resuscitation. 2023 Jul;188:109785. doi: 10.1016/j.resuscitation.2023.109785. Epub 2023 Apr 3. PMID 37019352
- [Background] Cocchi MN, Lucas JM, Salciccioli J, Carney E, Herman S, Zimetbaum P, Donnino MW. The role of cranial computed tomography in the immediate post-cardiac arrest period. Intern Emerg Med. 2010 Dec;5(6):533-8. doi: 10.1007/s11739-010-0403-8. Epub 2010 May 8. PMID 20454869
- [Background] Reynolds AS, Matthews E, Magid-Bernstein J, Rodriguez A, Park S, Claassen J, Agarwal S. Use of early head CT following out-of-hospital cardiopulmonary arrest. Resuscitation. 2017 Apr;113:124-127. doi: 10.1016/j.resuscitation.2016.12.018. Epub 2017 Jan 3. PMID 28057527